CLINICAL TRIAL: NCT06553807
Title: The Effect of Education Given to Women With Low Genital Self Image on Satisfaction With Genital Appearance and Quality of Sexual Life
Brief Title: Genital Self İmage and Satisfaction With Genital Appearance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zehra CAN, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023/5160
Record Dates: First submitted 2024-06-13; First posted 2024-08-14 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-08

CONDITIONS: Women
Keywords: Genital self-image; Satisfaction with genital appearance; Women; Quality of sexual life

STUDY DESIGN:
Intervention Model Description: An educational booklet will be prepared, and a three-week educational program will be conducted for the intervention group, with one topic covered each week. The training sessions will be held three days a week, and the women will be divided into groups. Since the sample size is planned to be 40 participants, the training sessions will be organized into three separate groups, with sessions held on three designated days of the week (Monday, Tuesday, and Wednesday).
  Before the study begins, women who meet the inclusion criteria and agree to participate will be briefed about the study's purpose and process in a designated private room at the FHC.
  The data will be collected face-to-face in a private room at the FHC by the researcher during the application dates. Each training session is planned to last an average of 30-45 minutes. At the beginning of the first session, participants will be given the educational booklet.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will consist of women who score 21 points or less on the Genital Self-Image Scale.
  Interventions: Other: The intervention group, which was randomly selected by randomisation and accepted to participate in the study, is planned to receive 3-week training sessions between 30-45 minutes.
- Control (No Intervention): The control group will consist of women who score 21 points or less on the Genital Self-Image Scale.

INTERVENTIONS:
Other: The intervention group, which was randomly selected by randomisation and accepted to participate in the study, is planned to receive 3-week training sessions between 30-45 minutes. — The intervention group, which was randomly selected by randomisation and accepted to participate in the study, is planned to receive 3-week training sessions between 30-45 minutes. Pre-test and post-test will be applied to the participants after 4 weeks. Follow-up test data will be collected from the intervention and control groups after 3 months.
  Arms: Intervention

SUMMARY:
The concept of genital self-image first emerged alongside genital identity. Womens perceptions of their genital self encompass their feelings and subjective thoughts about their sexual organs. One of the most significant problems resulting from a negative genital self-image is sexual health. It has been reported that genital self-perception and self-image are related to sexual health. Another study that examined the effects of viewing various vulvar photographs on womens genital attitudes found that women had relatively positive genital self-images before viewing the photographs, but their perceptions became even more positive after viewing them. This study aims to examine the impact of education on genital appearance satisfaction and sexual quality of life in women with low genital self-image. It is hypothesized that women with low genital self-image who receive education will have more knowledge about genital anatomy, which will positively influence their genital appearance, genital self-image, and consequently improve their sexual quality of life.

The study is a randomized controlled experimental research. The research will be conducted women aged 18-49 years with low genital self-image who are registered at a Family Health Center (FHC). Data collection tools in the study will include a socio-demographic data form prepared by the researchers, the Genital Self-Image Scale, the Genital Appearance Satisfaction Scale, and the Sexual Quality of Life Scale. The SPSS 24.0 software package is planned to be used for data analysis. Descriptive statistics such as mean, standard deviation, number, and percentage will be used in the analysis of the quantitative data. The normality of the data distribution will be assessed, and parametric or non-parametric tests will be applied based on the distribution. Additionally, regression analyses will be used to evaluate the effect, and a significance level of 0.05 will be accepted for the entire study.

DETAILED DESCRIPTION:
The concept of genital self-image first emerged alongside genital identity. Much of the research on self-image has focused on womens attitudes towards beauty, weight, and skin color, often excluding issues related to genital/vaginal self-image. Womens perceptions of their genital self encompass their feelings and subjective thoughts about their sexual organs. The appearance and function of the genital area form the basis of genital self-image for women. Many women lack knowledge about certain anatomical features of their genital area, which is often seen as a taboo subject. This taboo can lead to women perceiving their genital organs as foreigns or unknowns. Although women generally report moderately positive genital self-perceptions, many are dissatisfied with their sexual organs in general or with one or more aspects of them at some point in their lives.

One of the most significant problems resulting from a negative genital self-image is sexual health. It has been reported that genital self-perception and self-image are related to sexual health. Sexual quality of life, which is a component of overall quality of life, is generally defined as how satisfied an individual is with their sexual life. It is thought that satisfaction with genital appearance and genital self-image can affect sexual quality of life. One study found that an increase in genital self-image was associated with an increase in sexual quality of life. Another study discovered that genital self-image was strongly related to sexual functionality and satisfaction. In a different study, women with a negative genital self-image were found to have more body and genital self-consciousness, less sexual pleasure, lower sexual esteem, less sexual functionality, and fewer experiences with various sexual activities. The continuation of this taboo and the lack of knowledge about womens genital appearances can lead to numerous problems. It has been suggested that education aimed at addressing these knowledge gaps could improve perceptions of genital appearance. A study investigating the effectiveness of a video education on genital appearance found that it significantly improved womens perceptions and awareness of genital diversity and resulted in a small but significant decrease in genital appearance dissatisfaction. Another study that examined the effects of viewing various vulvar photographs on womens genital attitudes found that women had relatively positive genital self-images before viewing the photographs, but their perceptions became even more positive after viewing them.

This study aims to investigate the impact of education on genital appearance satisfaction and sexual quality of life in women with low genital self-image. It is hypothesized that women with low genital self-image who receive education will have more knowledge about genital anatomy, which will positively influence their genital appearance, genital self-image, and consequently improve their sexual quality of life.

1.1. Aim of the Study

Aim: This study aims to examine the impact of education on genital appearance satisfaction and sexual quality of life in women with low genital self-image.

Research Hypotheses:

H1a: The education provided to women with low genital self-image has no effect on genital appearance satisfaction.

H1b: The education provided to women with low genital self-image has an effect on genital appearance satisfaction.

H2a: The education provided to women with low genital self-image has no effect on sexual quality of life.

H2b: The education provided to women with low genital self-image has an effect on sexual quality of life.

Research Overview The study is a randomized controlled experimental research.

The research will be conducted on women aged 18-49 years with low genital self-image, registered at the Family Health Center (FHC) , Turkey. The research population consists of women registered at the FHC in the specified province. The sample includes women aged 18-49 years with low genital self-image determined by the Genital Self-Image Scale. The sample size will be determined using the Genital Self-Image Scale.

Based on a similar study, a Power analysis (G*Power 3.1) determined a minimum of 30 participants each for the intervention and control groups, totaling 60 participants, considering an effect size of 0.98, a 0.05 margin of error, and 0.05 significance. Given potential losses, the study plans to include 80 participants (40 in each group). Participants were assigned to intervention and control groups using simple randomization. The intervention group will receive a 3-week training session, with each session lasting 30-45 minutes.

Study Groups There will be two groups: control and intervention. Women scoring 21 or below on the Genital Self-Image Scale will form the groups. Participants were assigned to intervention and control groups using simple randomization with the http://biostatapps.inonu.edu.tr/RAY/ program. Data collection tools will include a socio-demographic data form prepared by the researchers, the Genital Self-Image Scale, the Genital Appearance Satisfaction Scale, and the Sexual Quality of Life Scale. Participants will be informed about the studys purpose and content, and those meeting the inclusion criteria will provide verbal and written informed consent.

Data Collection Pre-test data will be collected face-to-face at the FHC. Post-test data will be collected four weeks after the interventions for the intervention group and four weeks after the pre-test for the control group. Follow-up data will be collected three months later through face-to-face interviews.

Nursing Intervention

An educational booklet will be prepared, and training will be conducted over three weeks, with three sessions each week. The training sessions will cover:

1. Anatomy and physiology of the reproductive system, including sexual organs.
2. Normal genital appearance and changes in the genital area during different life stages (adolescence, fertility, menopause).
3. Information on genital appearance satisfaction and perceptions. Participants will be encouraged to ask questions. Post-training and three months later, participants will fill out the survey and scales again.

Intervention Group Women in the intervention group will receive three weeks of training sessions lasting 30-45 minutes each. The intervention group will complete pre-test scales before the training and post-test scales four weeks after the training.

Variables Dependent Variables: Scores from the Genital Appearance Satisfaction Scale, Genital Self-Image Scale, and Sexual Quality of Life Scale.

Independent Variable: The training provided to women with low genital self-image.

Control Variables: Characteristics such as age, education level, occupation, economic status, BMI, and smoking and alcohol use, as well as aspects related to sexual life.

Data Analysis Data analysis will use SPSS 24.0. Descriptive statistics such as mean, standard deviation, number, and percentage will be used. The normality of the data distribution will be assessed, and parametric or non-parametric tests will be applied accordingly. Cronbachs alpha coefficients will be calculated for the scales used. Differences between groups will be analyzed, and post hoc tests will be used if necessary. Regression analyses will evaluate the effect, with a significance level of 0.05 for the entire study.

Ethical Considerations Ethical approval was obtained from the İnönü University Non-Interventional Clinical Research and Publication Ethics Committee. Institutional permissions were also secured for conducting the research.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years old,
* Sexually active for at least 1 year,
* Not having language and communication problems,
* Literate.

Exclusion Criteria:

* Pregnancy within the last year,
* She had a previous gynaecological operation,
* Experiencing early menopause,
* Diagnosed with gynaecological cancer or undergoing cancer treatment,

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The research is planned to be applied only to women
Enrollment: 80 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
The Effect of Education Given to Women With Low Genital Self Image on Satisfaction With Genital Appearance and Quality of Sexual Life | 1 year
  Socio-demographic Data Form: Socio-demographic data form consists of a total of 12 questions.
  Genital Appearance Satisfaction Scale: It consists of 11 items related genital appearance. A minimum score of "0" and a maximum score of "33" can be obtained from scale. The higher score obtained from scale, higher dissatisfaction with genital appearance.
  Female Genital Self-Image Scale: It is a 7-item 4-point Likert-type scale that evaluates women's feelings and beliefs about their genitals. Scale scores range from 7 to 28, with higher scores indicating more favourable genital self-image.
  Sexual Quality of Life Scale-Female (CYKÖ-K): CYKÖ-K is six-point Likert-type and consists of 18 items. The range of points that can be obtained from scale in the 1-6 scoring is between 18-108. 0-5 scoring, score range is 0-90. A high score on the scale indicates that the quality of sexual life is good. The relationship and impact between the scores of the scales will be evaluated.

IPD SHARING:
Plan to Share IPD: No
data can be shared upon request